CLINICAL TRIAL: NCT01868763
Title: TeleLifestyleCoaching Use of Telemedicine for Weight Loss and Care of Weight Associated Illnesses
Brief Title: TeleLifestyleCoaching for Weight Loss
Acronym: FitMeFit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West German Center of Diabetes and Health (Other)
Collaborators: HMM Holding AG (Unknown)
Responsible Party: Principal Investigator, Stephan Martin, Director, West German Center of Diabetes and Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FitMeFit
Record Dates: First submitted 2013-05-30; First posted 2013-06-05 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: Overweight
Keywords: telemedicine; coaching; lifestyle change; weight loss
MeSH Terms: conditions — Overweight; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- control (C) group (No Intervention): The control group will remain in routine care for 12 weeks.
- telemedical (TM) group (Experimental): Participants in the telemedical (TM) group will get a weighing machine and a step counter, with automatic transfer into a personalized online portal, which can be monitored from both, the participant and the study centre.
  Interventions: Device: telemedical devices (weighing machine and step counter)
- telemedical coaching (TMC) group (Experimental): Participants in the telemedical coaching (TMC) group will get a weighing machine and a step counter, with automatic transfer into a personalized online portal, which can be monitored from both, the participant and the study centre. Additionally, they will be called once per week for 12 weeks from the study centre aiming to discuss measured data and to fix target agreements.
  Interventions: Device: telemedical devices (weighing machine and step counter); Behavioral: care calls once per week for 12 weeks

INTERVENTIONS:
Device: telemedical devices (weighing machine and step counter)
  Arms: telemedical (TM) group; telemedical coaching (TMC) group
Behavioral: care calls once per week for 12 weeks
  Arms: telemedical coaching (TMC) group

SUMMARY:
Lifestyle changes often fail due to loss of motivation. Telemedicine and personal coaching have the potential to support lifestyle change and weight loss. Therefore, the aim of our randomized controlled trial was to examine the effect of telemedicine with and without coaching in comparison to a control group on weight loss in overweight participants.

DETAILED DESCRIPTION:
In an occupational health care setting overweight employees were randomized into a three arm 12-week trial. Participants in the telemedical (TM) and telemedical coaching (TMC) group got a weighing machine and a step counter, with automatic transfer into a personalized online portal, which could be monitored from both, the participant and the study centre. The TMC group weekly got care calls from the study centre aiming to discuss measured data and to fix target agreements. The control group remained in routine care. Wilcoxon signed rank test was used to determine if differences (baseline vs. after 12 weeks) were significantly different from 0 and ANOVA test for determination of inter group differences.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥27 kg/m2

Exclusion Criteria:

* Hypoglycemia inducing medication
* severe disease with hospital stay during the last 3 months
* smoking cessation for less then 3 months
* planned smoking cessation during study phase
* acute infects
* chronic diseases

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2012-08; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
weight loss | 12 weeks
  Weight will be measured at baseline and after 12 weeks

SECONDARY OUTCOMES:
cardiometabolic risk factors | 12 weeks
  Body mass index [kg/m2], waist circumference [cm], blood pressure [mmHg], triglycerides [mg/dl], HbA1c [%], total, HDL and LDL cholesterol [mg/dl]

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Martin, MD, Principal Investigator — West-German Centre of Diabetes and Health
Locations (1):
- West-German Centre of Diabetes and Health, Düsseldorf, Germany

REFERENCES:
- [Derived] Kempf K, Rohling M, Stichert M, Fischer G, Boschem E, Konner J, Martin S. Telemedical Coaching Improves Long-Term Weight Loss in Overweight Persons: A Randomized Controlled Trial. Int J Telemed Appl. 2018 Sep 9;2018:7530602. doi: 10.1155/2018/7530602. eCollection 2018. PMID 30271433